CLINICAL TRIAL: NCT00166751
Title: Sonographic Assessment of Laryngeal Elevation in Cerebrovascular Accident Patients With Dysphagia
Brief Title: Sonographic Assessment of Laryngeal Elevation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701221
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2004-12

CONDITIONS: Cerebrovascular Accident; Dysphagia
Keywords: Videofluoroscopic examination,; ultrasound; laryngeal elevation; dysphagia
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Ultrasonographic examination has long been used to assess the swallowing function. It has the advantages of no ionizing radiation on examination and the possibility of using the real food instead of the barium meal in testing. Thus, the subjects can be examined repeatedly and in a more physiological status of swallowing. However, the ultrasonographic examination is only used in assessing the oral phase of swallowing. It can accurately visualize the tongue movement, measure the oral transit time of bolus, and sometimes the hypoid bone motion, but has not been applied on the evaluation of pharyngeal phase of swallowing. Physically, laryngeal elevation is an essential component of the swallowing movement on pharyngeal phase. It ensures the occlusion of airway and opening of criopharymgeus muscle, and thus prevents the aspiration. To evaluate the laryngeal elevation is crucial point in managing the dysphagic patients.

The purpose of this project is to measure the laryngeal elevation in normal and in dysphagic patients with cerebrovascular (CVA) accident using ultrasonographic techniques. This work will include four group subjects. The first group consists of 20 young subjects (< 40 years); the second group consists of 20 age-matched normal subjects; the third group consists of 20 CVA patients without swallowing problems, and the fourth group consists of 20 CVA patients with dysphagia, which was proven by VFSS. The laryngeal elevation is detected by ultrasound with the transducer placing between the hyoid bone and thyroid cartilage. The two markers are easily detected on sonogram because of the presence of acoustic shadow, a specific character of bony structure on sonogram. The distance between the hyoid bone and thyroid cartilage before and during swallowing is measures and compared among the groups. The distance change of the patients with dysphagia is further compared with that defined by VFSS. With the result of this study, we will understand the status of laryngeal elevation during swallowing in normal and dysphagic subjects, and further determine the accuracy of ultrasonographic measurement in measuring the laryngeal elevation. With this knowledge, we might extend the usage of ultrasonographic examination on evaluating swallowing function.

DETAILED DESCRIPTION:
Dysphagia is a common problem in rehabilitation medicine. To accurately evaluate its disorder is crucial in managing this group patient. Videofluoroscopic examination of swallow (VFSS) is generally regarded as the "gold standard" in the assessment of oropharyngeal dysphagia, especially in the detection of laryngeal penetration or subglottic aspiration. However, its limitations are widely acknowledged. VFSS cannot be performed widely because of its radiation exposure, is a single time measure, where as aspiration may be a variable phenomenon. Moreover, VFSS may over diagnose the disorder of swallowing function since the unflavored barium could disturb deglutition ability of the patients, particularly in those who having impaired cognitive function. As a result, the researchers have sought for more reliable bedside evaluation methods to detect aspiration. Various bedside clinical evaluations such as neurological examination, water swallow test, and swallowing provocation test have been used in identifying predicting or aspiration. However, when considered against the gold standard VFSS, prediction rate for aspiration was still unsatisfactory. Seeking for more non-invasive and objective method of evaluating swallowing function is continuing by many researches.

Ultrasonographic examination has long been used to assess the swallowing function. It has the advantages of no ionizing radiation on examination and the possibility of using the real food instead of the barium meal in testing. Thus, the subjects can be examined repeatedly and in a more physiological status of swallowing. However, the ultrasonographic examination is only used in assessing the oral phase of swallowing. It can accurately visualize the tongue movement, measure the oral transit time of bolus, and sometimes the hypoid bone motion, but has not been applied on the evaluation of pharyngeal phase of swallowing. Physically, laryngeal elevation is an essential component of the swallowing movement on pharyngeal phase. It ensures the occlusion of airway and opening of criopharymgeus muscle, and thus prevents the aspiration. To evaluate the laryngeal elevation is crucial point in managing the dysphagic patients.

The purpose of this project is to measure the laryngeal elevation in normal and in dysphagic patients with cerebrovascular (CVA) accident using ultrasonographic techniques. This work will include four group subjects. The first group consists of 20 young subjects (< 40 years); the second group consists of 20 age-matched normal subjects; the third group consists of 20 CVA patients without swallowing problems, and the fourth group consists of 20 CVA patients with dysphagia, which was proven by VFSS. The laryngeal elevation is detected by ultrasound with the transducer placing between the hyoid bone and thyroid cartilage. The two markers are easily detected on sonogram because of the presence of acoustic shadow, a specific character of bony structure on sonogram. The distance between the hyoid bone and thyroid cartilage before and during swallowing is measures and compared among the groups. The distance change of the patients with dysphagia is further compared with that defined by VFSS. With the result of this study, we will understand the status of laryngeal elevation during swallowing in normal and dysphagic subjects, and further determine the accuracy of ultrasonographic measurement in measuring the laryngeal elevation. With this knowledge, we might extend the usage of ultrasonographic examination on evaluating swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* 1.stroke with clear consciousness 2.Abnormal videofluoroscopic examination 3.Good cooperation

Exclusion Criteria:

* 1. Lung infection 2. Can not oral feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-09; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Tyng-Guey Wang, MD, Principal Investigator — National Taiwan University, School of Medicine, National Taiwan University
Locations (1):
- Tyng-Guey Wang, Taipei, Taiwan